CLINICAL TRIAL: NCT01032642
Title: A Simple Technique to Reduce the Pain in Hysterosalpingography Using A Thin Catheter
Brief Title: A Thin Catheter For Hystrosalpingography
Acronym: HSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: The Egyptian IVF-ET Center (Other)
Responsible Party: Ragaa Mansour, The Egyptian IVF-ET center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Inany-1
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2008-09

CONDITIONS: Infertility
Keywords: infertility fallopian tubes
MeSH Terms: conditions — Infertility | interventions — Hysterosalpingography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thin catheter group (Experimental): group of women where thin catheter will be used for hysterosalpingography
  Interventions: Device: device for hysterosalpingography

INTERVENTIONS:
Device: device for hysterosalpingography — a thin catheter originally designed for IUI (sperm processor cat. No. SP/PL/01, Aurangabad, India) connected to a 10 mL syringe filled with urographin 76% (Scherring, Germany) will be introduced through the cervical canal into the lower part of the uterine cavity. After introducing the catheter, the screw of the vaginal speculum will be loosened to allow the two valves of the speculum to press on the portiovaginalis of the cervix to prevent leakage of the dye. Then the dye will be injected slowly and the procedure will be watched on the screen and x-ray films will be taken.

SUMMARY:
The investigators will use a thin catheter for HSG and apply pressure on the cervix with the vaginal speculum to prevent leakage of the dye during injection to study the uterine cavity and fallopian tubes and reduce the pain as compared to a standard metal cannula.

DETAILED DESCRIPTION:
Hysterosalpingography (HSG) remains one of the most reliable methods to study tubal patency and the uterine cavity (1-3). The relative indications and importance of HSG and laparoscopy in the diagnosis of tubal factor infertility have been extensively discussed. Recently a multicenter randomized controlled trial (4) has demonstrated that the routine use of HSG at an early stage of infertility work up, prior to laparoscopy and dye, does not influence the cumulative pregnancy rate compared with the routine use of laparoscopy and dye alone. However, HSG is an efficient method which is less invasive and less costly than laparoscopy (5), and than transvaginal hydrolaparoscopy (6). The main disadvantages of HSG are being unable to confirm adhesions, endometriosis and being a painful procedure (7,8). Different cannulas and catheters have been tried to reduce pain such as the Rubin cannula (9), Jorcho cannula (10), and Whitehead cannula or Foley catheter (11). Minimal difference in the degree of pain was found when the balloon catheter was compared with the cervical cup (12). General and local medications have been tried to alleviate pain during the procedure. (3,13).

HSG is widely practiced in our country, however, for cost effective reasons, the standard metal cannula is the only method used at our hospital. It is painful procedure because it requires grasping the cervix with a tenaculum and inducing some cervical dilatation during introduction of the cannula. The aim of this pilot study was to develop a simple and painless technique for HSG using a thinner than normal catheter, and without grasping the cervix with a tenaculum. Leakage of the dye through the cervix was prevented by pressing on the portiovaginalis of the cervix using the vaginal speculum. This technique for performing HSG is a novel one and has not been described previously in the medical literature.

ELIGIBILITY:
Inclusion Criteria:

* infertile women during their fertility workup and requesting to do hysterosalpingography

Exclusion Criteria:

* women with pelvic inflammatory disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
pain score during introduction of catheter and during the injection of dye | 3-6 month
the efficiency of the new technique in filling the uterine cavity with the dye and studying fallopian tubes | 3-6 month

SECONDARY OUTCOMES:
adverse events | within the study period

CONTACTS AND LOCATIONS:
Overall Officials: ragaa mansour, PhD, Principal Investigator — Egyptian IVF Center; hesham Al-Inany, PhD, Study Director — Kasr Al-Aini Hospital
Locations (1):
- kasr Al-Aini hospital, Cairo, Cairo Governorate, Egypt